CLINICAL TRIAL: NCT02110524
Title: Prospective, Controlled, Multi-Center, Open, Single Arm Study for the Treatment of Subjects Presenting De Novo Occluded/Stenotic or Re-occluded/Restenotic Lesions of the Superficial Femoral or Popliteal Arteries Using a Paclitaxel-Coated Percutaneous Angioplasty Catheter
Brief Title: CVI Drug Coated Balloon First In Human Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spectranetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP1027
Record Dates: First submitted 2014-04-04; First posted 2014-04-10 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Peripheral Arterial Disease
Keywords: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Angioplasty; Catheters

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CVI Drug Coated Balloon (Experimental)
  Interventions: Device: Percutaneous Transluminal Angioplasty

INTERVENTIONS:
Device: Percutaneous Transluminal Angioplasty
  Other Names: CVI Paclitaxel-coated, Percutaneous Transluminal Angioplasty (PTA) Balloon; Catheter

SUMMARY:
The purpose of this study is to assess safety and the inhibition of restenosis of the CVI Paclitaxel-coated PTA Balloon Catheter in the treatment of de-novo occluded/stenotic or reoccluded/restenotic superficial femoral (SFA) or popliteal arteries.

The primary endpoint for this analysis is late lumen loss at six (6) months.

DETAILED DESCRIPTION:
Prospective, controlled, multi-center, open, single arm study

Main cohort: 50; pre-specified treatment group: 30. Total patients: 80

ELIGIBILITY:
Inclusion Criteria:

* Subjects with symptomatic leg ischemia, requiring treatment of SFA or popliteal (P1 segment) artery
* De novo or restenotic lesion(s) >70% within the SFA and popliteal arteries in a single limb which are ≥3 cm and ≤15 cm in cumulative total length (by visual estimation).
* Target vessel reference diameter ≥3 mm and ≤7 mm (by visual estimation).
* Rutherford classification of 2, 3 or 4

Exclusion Criteria:

* Lesion length is <3 cm or >15 cm or there is no normal proximal arterial segment in which duplex ultrasound velocity ratios can be measured.
* Outflow arteries (distal popliteal, anterior or posterior tibial or peroneal arteries) with significant lesions (≥ 50% stenosis) may not be treated during the same procedure.
* Treatment of the contralateral limb during the same procedure or within 30 days of the study procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-12; Primary Completion 2012-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Primary endpoint: Angiographic late lumen loss | 6Month
  difference between minimum lumen diameter after intervention and follow up.

SECONDARY OUTCOMES:
Secondary safety endpoint: Major Adverse Event (MAE) rate | 6Months
  composite rate of cardiovascular death, index limb amputation and ischemia driven target lesion revascularization (TLR).

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Schröder, MD, Principal Investigator — Jewish Hospital Berlin
Locations (1):
- Jewish Hospital Berlin, Berlin, Germany

REFERENCES:
- [Derived] Gray WA, Jaff MR, Parikh SA, Ansel GM, Brodmann M, Krishnan P, Razavi MK, Vermassen F, Zeller T, White R, Ouriel K, Adelman MA, Lyden SP. Mortality Assessment of Paclitaxel-Coated Balloons: Patient-Level Meta-Analysis of the ILLUMENATE Clinical Program at 3 Years. Circulation. 2019 Oct;140(14):1145-1155. doi: 10.1161/CIRCULATIONAHA.119.040518. Epub 2019 Sep 30. PMID 31567024